CLINICAL TRIAL: NCT05568043
Title: The Reducing Respiratory Emergency Visits Using Implementation Science Interventions Tailored to Setting (REVISITS) Study: A Cluster Randomized Trial
Brief Title: The Reducing REVISITS Study: A Cluster RCT
Acronym: REVISITS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Society of Hospital Medicine (Other); Onda Collective (Unknown); The Hospital Medicine Reengineering Network (HOMERuN) (Unknown); COPD Foundation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 20-0373; 5R01HL146644-05 (NIH)
Record Dates: First submitted 2022-07-14; First posted 2022-10-05 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: COPD; COPD Exacerbation Acute
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: 2x2 with 2 intervention delivery methods (virtual vs. in-person) and 2 implementation support mechanisms (virtual mentoring vs. virtual mentoring plus co-design)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- In-person intervention delivery with virtual mentoring (Experimental): The implemented interventions will be in-person and will include virtual mentoring. The mentored implementation model (MIM) is an evidence-based strategy to promote the success and sustainability of hospital-based quality improvement (QI) initiatives. After completing the contextual assessments and pre-implementation planning in Aim 1, the investigators will collaborate with the SHM to harness their expertise with the MIM to implement the COPD Program over a one-year period during Aim 2 (implementation). Virtual Mentored Implementation involves implementing their assigned care transition program intervention delivery method using an innovative virtual mentored implementation approach using tele-conferencing technology (i.e., video-conferences) for two-way visualization of individuals in different locations for educational purposes. Monthly mentoring sessions will occur to maximize mentors' input.
  Interventions: Behavioral: COPD Transitions of Care Intervention Bundle: In-Person Interventions
- In-person intervention delivery with virtual mentoring and co-design (Experimental): The implemented interventions will be in-person and will include virtual mentoring and co-design support with our study partner, Onda Collective. The mentored implementation model (MIM) is an evidence-based strategy to promote the success and sustainability of hospital-based quality improvement (QI) initiatives. After completing the contextual assessments and pre-implementation planning in Aim 1, the investigators will collaborate with the SHM to harness their expertise with the MIM to implement the COPD Program over a one-year period during Aim 2 (implementation). Virtual Mentored Implementation involves implementing their assigned care transition program intervention delivery method using an innovative virtual mentored implementation approach using tele-conferencing technology (i.e., video-conferences) for two-way visualization of individuals in different locations for educational purposes. Monthly mentoring sessions will occur to maximize mentors' input.
  Interventions: Behavioral: COPD Transitions of Care Intervention Bundle: In-Person Interventions
- Virtual intervention delivery with virtual mentoring (Experimental): The implemented interventions will be virtual and will include virtual mentoring. The mentored implementation model (MIM) is an evidence-based strategy to promote the success and sustainability of hospital-based quality improvement (QI) initiatives. After completing the contextual assessments and pre-implementation planning in Aim 1, the investigators will collaborate with the SHM to harness their expertise with the MIM to implement the COPD Program over a one-year period during Aim 2 (implementation). Virtual Mentored Implementation involves implementing their assigned care transition program intervention delivery method using an innovative virtual mentored implementation approach using tele-conferencing technology (i.e., video-conferences) for two-way visualization of individuals in different locations for educational purposes. Monthly mentoring sessions will occur to maximize mentors' input.
  Interventions: Behavioral: COPD Transitions of Care Intervention Bundle: Virtual Interventions
- Virtual intervention delivery with virtual mentoring with co-design (Experimental): The implemented interventions will be virtual and will include virtual mentoring and co-design support with our study partner, Onda Collective. The mentored implementation model (MIM) is an evidence-based strategy to promote the success and sustainability of hospital-based quality improvement (QI) initiatives. After completing the contextual assessments and pre-implementation planning in Aim 1, the investigators will collaborate with the SHM to harness their expertise with the MIM to implement the COPD Program over a one-year period during Aim 2 (implementation). Virtual Mentored Implementation involves implementing their assigned care transition program intervention delivery method using an innovative virtual mentored implementation approach using tele-conferencing technology (i.e., video-conferences) for two-way visualization of individuals in different locations for educational purposes. Monthly mentoring sessions will occur to maximize mentors' input.
  Interventions: Behavioral: COPD Transitions of Care Intervention Bundle: Virtual Interventions

INTERVENTIONS:
Behavioral: COPD Transitions of Care Intervention Bundle: Virtual Interventions — The COPD Transitions of Care Intervention Bundle will be site-specific determined through Aim 1 contextual assessments and will consist of 2-3 evidence-based COPD transitions of care interventions. Virtual interventions included in the bundle may consist of: phone or e-consults for medication reconciliation, virtual teach-to-goal [V-TTG] or tele-TTG inhaler education, and post-discharge phone call communication and/or texts/ and/or electronic portal use, among others.
  Other Names: COPD Transitions of Care Program: Virtual Interventions
  Arms: Virtual intervention delivery with virtual mentoring; Virtual intervention delivery with virtual mentoring with co-design
Behavioral: COPD Transitions of Care Intervention Bundle: In-Person Interventions — The COPD Transitions of Care Intervention Bundle will be site-specific determined through Aim 1 contextual assessments and will consist of 2-3 evidence-based COPD transitions of care interventions. In-person interventions include face-to-face general COPD education, inhaler education, medication reconciliation, post-discharge clinic visits, community health worker home visits, pulmonary rehabilitation, smoking cessation programs, among others.
  Other Names: COPD Transitions of Care Program: In-Person Interventions
  Arms: In-person intervention delivery with virtual mentoring; In-person intervention delivery with virtual mentoring and co-design

SUMMARY:
This type II hybrid effectiveness-implementation trial will concurrently study the comparative effectiveness of virtual vs. in-person COPD care transition programs implemented via virtual mentored implementation approaches with and without co-design methods.

The investigators will enroll up to 24 randomized sites (with a goal minimum of 16 sites) to:

* Deliver the COPD programs implemented via mentored support in collaboration with SHM Center for Quality Improvement.
* Compare the effectiveness and penetration of virtual versus in-person COPD care transition programs implemented along with mentoring support with or without co-design.

The investigators aim to determine which combined approach(es) is/are the most effective at implementing evidence-based COPD program interventions and decreasing COPD acute care revisits with the greatest overall impact and sustainability.

DETAILED DESCRIPTION:
The COPD programs will be implemented via mentored support in collaboration with the SHM Center for Quality Improvement. Up to twenty-four hospitals will be randomized to one of four dyads: 1) in-person intervention delivery with virtual mentoring; 2) 1) in-person intervention delivery with virtual mentoring and co-design; 3) virtual intervention delivery with virtual mentoring; or 4) virtual intervention delivery with virtual mentoring with co-design. The research will use a pragmatic type II hybrid effectiveness-implementation cluster randomized trial such that once the hospital is randomized, the assigned program delivery (virtual vs. in-person) will be implemented via their assigned mentoring approach (virtual mentoring with/without co-desig) using quality improvement efforts. Each hospital will work with their mentors to implement their COPD care transition program (bundle of 2-3 interventions) based on their site-specific implementation plan developed in Aim 1 (already approved under this IRB number) according to their assigned delivery (in-person vs. virtual) over a one-year period; half of sites will also receive co-design support.

The mentored implementation model (MIM) is an evidence-based strategy to promote the success and sustainability of hospital-based quality improvement (QI) initiatives. After completing the contextual assessments and pre-implementation planning in Aim 1, the investigators will collaborate with the SHM to harness their expertise with the MIM to implement the COPD Program over a one-year period during Aim 2 (implementation). Virtual Mentored Implementation involves implementing their assigned care transition program intervention delivery method using an innovative virtual mentored implementation approach using tele-conferencing technology (i.e., video-conferences) for two-way visualization of individuals in different locations for educational purposes. In our proposal, the virtual site visits (≥1) and monthly mentoring sessions will use tele-conferencing so both the site-leads and mentor can visualize each other and the mentor can visualize and observe the site's additional team members, administrators, clinical and administrative space, data collection tools and technology, and any other resources and facilities that will allow the mentor to advise on optimal approaches for program implementation. Monthly mentoring sessions will occur using similar virtual teleconferencing technology to maximize mentors' input. Half of sites will also be randomized to co-design support with our study partner Onda Collective; the other half will only receive the virtual mentored support.

The sustainability of intervention and implementation outcomes will be evaluated at 6, 12, 18, and 24-months post-implementation. Mechanisms, moderators, and mediators will identify aspects of successful implementation, and program costs and savings will be analyzed across sites. These data will inform a dissemination strategy (e.g., toolkit) and will inform future large-scale implementation and cost-effectiveness studies. Site Leads will submit quarterly reports via REDCap and will be de-identified.

Qualitative contextual analyses across stakeholders (patients, clinicians, administrators) will assess for mediators, moderators, and mechanism of change using CFIR rating rules to determine valence (positive or negative influence on implementation and strength [influence on implementation weak or strong]). The investigators will use the CFIR matrix to compare within and across the up to 24 hospitals across each time point including baseline data collected in this context assessment, throughout relevant implementation time points, and post-implementation time points. To analyze the aggregate data, the investigators will use consensus-based coding: our team analysts will determine a summary rating using all of the individual, supporting qualitative, and rationale data into consideration and will discuss until the investigators reach consensus. Program costs/savings: The investigators will assess the value of implementation from the hospital's perspective, consistent with the study's focus on hospital-level implementation using implementation science economic evaluation principles to evaluate both the comparative program intervention and implementation costs. Principles of "cost of care" measures include actual costs (not billed costs), time-driven activity-based costing, and actual use of resources (actual time per patient, capacity cost, supporting costs), measured around the patient; implementation costs include: 1) startup costs: mentor training and education materials; 2) personnel costs (clinician/staff time); 3) supplies and space costs. The investigators will use monthly log sheets to collect the staff time and use self-administered tool to estimate startup costs. To calculate the costs of staff time, the investigators will determine an hourly wage on the basis of annual salaries and a 40-hour work week. All costs will be itemized and summarized annually with descriptive statistics including mean, SD, median, and interquartile range. To assess potential savings, value may be assessed differently depending on the sites' payment models. For instance, at sites that primarily or solely deliver care in fee-for-service payment models, reducing revisits may improve the quality of care, but not their financial bottom line, unless they significantly reduce their penalties under Medicare's HRRP. On the other hand, hospitals enrolled in value-based contracts, such as accountable care organizations and/or BPCI programs, may find that they are able to demonstrate improved savings or relative cost-savings by implementing programs. To determine overall value, the investigators will estimate site-specific 'savings' through estimated decreased Medicare penalties for excessive 30-day readmissions or by remaining under target for value-based purchasing contracts.

ELIGIBILITY:
Since enrollment for Aim 2 will occur on a site/system-level, the inclusion of specific individuals who meet these criteria are not applicable since Aim 2 will only enroll hospital sites, not individuals. The sites the investigators enroll will represent diverse patient populations and geographical locations across the US.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Healthcare Utilization: 30-day acute care revisits for COPD | Immediately Post-Program Implementation (12 months after enrollment in Aim 2)
  Composite of all emergency department visits and/or re-hospitalizations within 30-days post index hospitalization across all enrolled sites for COPD
Delivery of overall care transition program: penetration | Immediately Post-Intervention (12 months after enrollment in Aim 2)
  Proportion of hospitalized patients with COPD receiving their assigned care transition program interventions (composite) as per documented in the electronic health record.
Sustainability of effectiveness: 30-day revisits | Quarterly for 24 months Post-Intervention initial enrollment (Aim 3)
  Composite of all emergency department visits and/or re-hospitalizations within 30-days post index hospitalization.
Sustainability of program delivery: penetration | Quarterly for 24 months Post-Intervention initial enrollment (Aim 3)
  Proportion of hospitalized patients with COPD receiving their assigned care transition program interventions (composite) as per documented in the electronic health record.

SECONDARY OUTCOMES:
Delivery of care transition program individual interventions: penetration | Immediately Post-Intervention (12 months after enrollment in Aim 2)
  Proportion of patients with documented individual care transition interventions including: on admission and/or upon discharge medication reconciliation [yes/no]; self-management education, e.g., inhaler technique including baseline and/or post-education technique documentation [scores/descriptive] and/or whether education was provided [yes/no]; documentation that post-discharge communication occurred (Y/N); other site-specific care transition interventions (site-specific).
Cost/savings evaluation | At completion of 12- months of Intervention (Aim 3)
  To evaluate hospital-level program costs and savings.
Cost/savings evaluation | At 24 months Post-Intervention (Aim 3)
  To evaluate hospital-level program costs and savings.
Healthcare Utilization: 30-day acute care revisits for COPD during intervention | Immediately Post-Program Implementation (12 months after enrollment in Aim 2)
  Composite of all emergency department visits and/or re-hospitalizations within 30-days for COPD post index hospitalization across all enrolled sites.
Healthcare Utilization: 30-day acute care revisits for COPD | Post-Program Implementation (24 months after enrollment in Aim 3)
  Composite of all emergency department visits and/or re-hospitalizations within 30-days for COPD post index hospitalization across all enrolled sites.
Healthcare Utilization: 60-day acute care revisits for COPD | Immediately Post-Program Implementation (12 months after enrollment in Aim 2)
  Composite of all emergency department visits and/or re-hospitalizations within 60-days for COPD post index hospitalization across all enrolled sites.
Healthcare Utilization: 60-day acute care revisits for COPD | Post-Program Implementation (24 months after enrollment in Aim 3)
  Composite of all emergency department visits and/or re-hospitalizations within 60-days for COPD post index hospitalization across all enrolled sites.
Healthcare Utilization: 90-day acute care revisits for COPD | Immediately Post-Program Implementation (12 months after enrollment in Aim 2)
  Composite of all emergency department visits and/or re-hospitalizations within 90-days for COPD post index hospitalization across all enrolled sites.
Healthcare Utilization: 90-day acute care revisits for COPD | Post-Program Implementation (24 months after enrollment in Aim 3)
  Composite of all emergency department visits and/or re-hospitalizations within 90-days for COPD post index hospitalization across all enrolled sites.
Healthcare Utilization: 30-day acute care revisits (all cause) | Immediately Post-Program Implementation (12 months after enrollment in Aim 2)
  Composite of all emergency department visits and/or re-hospitalizations within 30-days post index hospitalization across all enrolled sites.
Healthcare Utilization: 30-day acute care revisits (all cause) | Post-Program Implementation (24 months after enrollment in Aim 3)
  Composite of all emergency department visits and/or re-hospitalizations within 30-days post index hospitalization across all enrolled sites.
Healthcare Utilization: 60-day acute care revisits (all cause) | Immediately Post-Program Implementation (12 months after enrollment in Aim 2)
  Composite of all emergency department visits and/or re-hospitalizations within 60-days post index hospitalization across all enrolled sites.
Healthcare Utilization: 60-day acute care revisits (all cause) | Post-Program Implementation (24 months after enrollment in Aim 3)
  Composite of all emergency department visits and/or re-hospitalizations within 60-days post index hospitalization across all enrolled sites.
Healthcare Utilization: 90-day acute care revisits (all cause) | Immediately Post-Program Implementation (12 months after enrollment in Aim 2)
  Composite of all emergency department visits and/or re-hospitalizations within 90-days post index hospitalization across all enrolled sites.
Healthcare Utilization: 90-day acute care revisits (all cause) | Post-Program Implementation (24 months after enrollment in Aim 3)
  Composite of all emergency department visits and/or re-hospitalizations within 90-days post index hospitalization across all enrolled sites.
Healthcare Utilization: 30-day emergency department revisits for COPD | Immediately Post-Program Implementation (12 months after enrollment in Aim 2)
  All emergency department visits within 30-days post index hospitalization for COPD across all enrolled sites.
Healthcare Utilization: 30-day emergency department revisits for COPD | Post-Program Implementation (24 months after enrollment in Aim 3)
  All emergency department visits within 30-days post index hospitalization for COPD across all enrolled sites.
Healthcare Utilization: 60-day emergency department revisits for COPD | Immediately Post-Program Implementation (12 months after enrollment in Aim 2)
  All emergency department visits within 60-days post index hospitalization for COPD across all enrolled sites.
Healthcare Utilization: 60-day emergency department revisits for COPD | Post-Program Implementation (24 months after enrollment in Aim 3)
  All emergency department visits within 60-days post index hospitalization for COPD across all enrolled sites.
Healthcare Utilization: 90-day emergency department revisits for COPD | Immediately Post-Program Implementation (12 months after enrollment in Aim 2)
  All emergency department visits within 90-days post index hospitalization for COPD across all enrolled sites.
Healthcare Utilization: 90-day emergency department revisits for COPD | Post-Program Implementation (24 months after enrollment in Aim 3)
  All emergency department visits within 90-days post index hospitalization for COPD across all enrolled sites.
Healthcare Utilization: 30-day emergency department revisits (all cause) | Immediately Post-Program Implementation (12 months after enrollment in Aim 2)
  All emergency department visits within 30-days post index hospitalization across all enrolled sites.
Healthcare Utilization: 30-day emergency department revisits (all cause) | Post-Program Implementation (24 months after enrollment in Aim 3)
  All emergency department visits within 30-days post index hospitalization across all enrolled sites.
Healthcare Utilization: 60-day emergency department revisits (all cause) | Immediately Post-Program Implementation (12 months after enrollment in Aim 2)
  All emergency department visits within 60-days post index hospitalization across all enrolled sites.
Healthcare Utilization: 60-day emergency department revisits (all cause) | Post-Program Implementation (24 months after enrollment in Aim 3)
  All emergency department visits within 60-days post index hospitalization across all enrolled sites.
Healthcare Utilization: 90-day emergency department revisits (all cause) | Immediately Post-Program Implementation (12 months after enrollment in Aim 2)
  All emergency department visits within 90-days post index hospitalization across all enrolled sites.
Healthcare Utilization: 90-day emergency department revisits (all cause) | Post-Program Implementation (24 months after enrollment in Aim 3)
  All emergency department visits within 90-days post index hospitalization across all enrolled sites.
Healthcare Utilization: 30-day re-hospitalizations for COPD | Immediately Post-Program Implementation (12 months after enrollment in Aim 2)
  All re-hospitalizations within 30-days post index hospitalization for COPD across all enrolled sites.
Healthcare Utilization: 30-day re-hospitalizations for COPD | Post-Program Implementation (24 months after enrollment in Aim 3)
  All re-hospitalizations within 30-days post index hospitalization for COPD across all enrolled sites.
Healthcare Utilization: 60-day re-hospitalizations for COPD | Immediately Post-Program Implementation (12 months after enrollment in Aim 2)
  All re-hospitalizations within 60-days post index hospitalization for COPD across all enrolled sites.
Healthcare Utilization: 60-day re-hospitalizations for COPD | Post-Program Implementation (24 months after enrollment in Aim 3)
  All re-hospitalizations within 60-days post index hospitalization for COPD across all enrolled sites.
Healthcare Utilization: 90-day re-hospitalizations for COPD | Immediately Post-Program Implementation (12 months after enrollment in Aim 2)
  All re-hospitalizations within 90-days post index hospitalization for COPD across all enrolled sites.
Healthcare Utilization: 90-day re-hospitalizations for COPD | Post-Program Implementation (24 months after enrollment in Aim 3)
  All re-hospitalizations within 90-days post index hospitalization for COPD across all enrolled sites.
Healthcare Utilization: 30-day re-hospitalizations (all cause) | Immediately Post-Program Implementation (12 months after enrollment in Aim 2)
  All re-hospitalizations within 30-days post index hospitalization across all enrolled sites.
Healthcare Utilization: 30-day re-hospitalizations (all cause) | Post-Program Implementation (24 months after enrollment in Aim 3)
  All re-hospitalizations within 30-days post index hospitalization across all enrolled sites.
Healthcare Utilization: 60-day re-hospitalizations (all cause) | Immediately Post-Program Implementation (12 months after enrollment in Aim 2)
  All re-hospitalizations within 60-days post index hospitalization across all enrolled sites.
Healthcare Utilization: 60-day re-hospitalizations (all cause) | Post-Program Implementation (24 months after enrollment in Aim 3)
  All re-hospitalizations within 60-days post index hospitalization across all enrolled sites.
Healthcare Utilization: 90-day re-hospitalizations (all cause) | Immediately Post-Program Implementation (12 months after enrollment in Aim 2)
  All re-hospitalizations within 90-days post index hospitalization across all enrolled sites.
Healthcare Utilization: 90-day re-hospitalizations (all cause) | Post-Program Implementation (24 months after enrollment in Aim 3)
  All re-hospitalizations within 90-days post index hospitalization across all enrolled sites.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Press, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee CT, Traeger L, Akula M, Fegley AE, Goldstein J, Erwin K, Damschroder LJ, Rommes J, Pick H, Auerbach A, Lindenauer P, Wan W, Jackson Sagredo A, Press VG. Virtual Mentored Implementation to Improve Care Transitions in Chronic Obstructive Pulmonary Disease: Protocol for a Pragmatic Implementation Study. JMIR Res Protoc. 2026 Jan 13;15:e82043. doi: 10.2196/82043. PMID 41529255